CLINICAL TRIAL: NCT06604039
Title: A Prospective Clinical Registry Evaluating Safety and Performance of Teleflex Vascular Access Devices
Brief Title: A Clinical Registry to Demonstrate the Safety and Performance of Teleflex Vascular Access Devices
Acronym: VADER
Status: Recruiting | Type: Observational
Sponsor: Teleflex (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-02
Record Dates: First submitted 2024-08-08; First posted 2024-09-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-09

CONDITIONS: Vascular Access Device
MeSH Terms: interventions — Central Venous Catheters; Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject: Needing a vascular access device for therapy or diagnosis
  Interventions: Device: Central venous catheter

INTERVENTIONS:
Device: Central venous catheter — Placement of a medical device to gain entry into the bloodstream, typically through a vein or artery, for the purpose of administering fluids, medications, blood products, or for hemodialysis
  Other Names: Peripherally inserted central catheter; Dialysis catheter; Midline intravenous catheter; Peripheral intravenous catheter; Arterial catheter; Catheter navigation/tip confirmation device

SUMMARY:
The general objective of Teleflex's Vascular Access Device Registry (VADER) is to provide high-quality Level 3 (or better) data on the performance, safety and clinical benefits of Teleflex's vascular access devices when used in a real-world setting

DETAILED DESCRIPTION:
The primary objective is to provide high-quality Level 3 (or better), data as defined by Medical Device Coordination group (MDCG) 2020-6, on the performance, and clinical benefits of Teleflex's vascular access devices when used in a real-world setting. The hypothesis is that, when used in accordance with the instructions for use (IFU), the vascular access devices will perform safely and successfully.

The Teleflex vascular access devices (index devices and accessories) in scope for this Registry vary in type from central venous access devices (CVAD) to midline catheters to peripheral catheters to hemodialysis catheters to arterial catheters navigation/tip confirmation devices. Many, but not all, of the devices also have antimicrobial and antithrombogenic properties. Also in scope are the accessories routinely used for placement and maintenance of the index devices.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will undergo a procedure that will include use of a Teleflex device covered by this Research.
* Subject is willing and capable of providing informed consent and/or give approval to collect, store and process limited health information by the Sponsor; or such consent is provided by a legally designated representative if required by local law or regulation.
* Subjects is able to read and understand English or Spanish languages

Exclusion Criteria:

* Subject is currently participating in another clinical Registry or investigation that may confound the results of this Registry.
* Subject was previously failed screening or was enrolled in this clinical Registry.
* Subject is imprisoned
* Subject is cognitively impaired and unable to provide informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who are scheduled to receive a vascular access procedure using at least one Teleflex vascular access device will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-12-08 (Actual); Primary Completion 2034-12-07 (Estimated); Study Completion 2034-12-07 (Estimated)

PRIMARY OUTCOMES:
Catheter devices: successful use of the device without removal due to device-related adverse events | Within 7 days after subject device removal
  The proportion of device uses successfully completed without device removal due to device-related adverse events
Arrow VPS Rhythm DXL catheter tip positioning system: Successful verification of catheter tip location | Immediately after subject device removal
  Successful verification of catheter tip location

SECONDARY OUTCOMES:
Device-related adverse events | Within 7 days after subject device removal
  Incidence of device-related adverse events during placement or use
Device-related adverse events within 7 days of device removal | Within 7 days after subject device removal
  Incidence of device-related adverse events following removal

OTHER OUTCOMES:
Adverse event caused by use of device accessory | Within 7 days after subject device removal
  Clinicians used accessory safely
Device accessory used successfully | Within 7 days after subject device removal
  Clinician used accessory successfully
Duration of use | Within 7 days after subject device removal
  How long the device was in use for the patient
Usability score | Within 7 days after subject device removal
  Subject device usability score. Medical Device Usability Score: Scale of 1-5 in which 1=very difficult, 2=difficult, 3=acceptable, 4=easy, 5=very easy

CONTACTS AND LOCATIONS:
Overall Officials: Amy Bardin, Study Director — Teleflex Incorporated Clinical and Medical Affairs
Locations (3):
- United States (3):
  - Huntsville Hospital, Huntsville, Alabama
  - Loma Linda University Health, Loma Linda, California
  - Tufts Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time